CLINICAL TRIAL: NCT01304069
Title: Effect of Celecoxib and Etoricoxib on the Pharmacokinetics and Pharmacodynamics of Oral Tramadol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Klaus T Olkkola, MD, Prof, Turku University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 119/180/2010; 2010-023373-19 (EudraCT Number)
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-07

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacodynamics
MeSH Terms: interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Selecoxib (Active Comparator)
  Interventions: Drug: Selecoxib
- Etoricoxib (Active Comparator)
  Interventions: Drug: Etoricoxib

INTERVENTIONS:
Drug: Placebo — The subjects will be given orally placebo twice a day for 7 days prior to the study.
  Arms: Placebo
Drug: Selecoxib — The subjects will be given orally selecoxib 200mg twice a day for 7 days prior to the study.
  Arms: Selecoxib
Drug: Etoricoxib — The subjects will be given orally etoricoxib 120mg once a day for 7 days prior to the study.
  Arms: Etoricoxib

SUMMARY:
Tramadol is an opioid analgesic, which is widely used in the treatment of acute and neuropathic pain. After oral administration, tramadol is rapidly and almost completely absorbed. Tramadol is extensively metabolised by O- and N-demethylation, which are catalysed by the liver CYP-450 enzymes. O-desmethyltramadol is an active metabolite and its formation is catalysed by CYP2D6. This study is aimed to investigate the possible interaction of oral tramadol with selecoxib and etoricoxib. Selecoxib is known to inhibit CYP2D6. Twelve healthy male or female adult non-smoking volunteers aged 18-40 years with body weights within ±15% of the ideal weight for height are taken into the study. Primary endpoints of the study are plasma concentrations of tramadol and its metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 18-40
* Body weight within ±15% of the ideal weight for height

Exclusion Criteria:

* A previous history of intolerance to the study drugs or to related compounds and additives
* Concomitant drug therapy of any kind for at least 14 days prior to the study
* Existing or recent significant disease
* History of hematological, endocrine, metabolic or gastrointestinal disease, including gut motility disorders
* History of asthma or any kind of drug allergy
* Previous or present alcoholism, drug abuse, psychological or other emotional problems that are likely to invalidate informed consent, or limit the ability of the subject to comply with the protocol requirements
* A positive test result for urine toxicology
* A "yes" answer to any one of the Abuse Questions
* Pregnancy or nursing
* Donation of blood for 4 weeks prior and during the study
* Special diet or life style conditions which would compromise the conditions of the study or interpretation of the results
* Participation in any other studies involving investigational or marketed drug products concomitantly or within one month prior to the entry into this study
* Smoking for one month before the start of the study and during the whole study period
* Any history of coagulation abnormality, also in first degree relatives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Concentration of tramadol and its metabolites in plasma | 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours after administration of tramadol

SECONDARY OUTCOMES:
Serotonin concentrations | 0, 4 and 8 hours after tramadol administration
  Serotonin concentrations will be analyzed with chromatographical methods from the blood samples drawn 0, 4 and 8 hours after tramadol administration
Pharmacodynamic effects | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after administration of tramadol
  The psychomotor effects of tramadol will be assessed with the measurement of pupil size with Cogan's pupillometer, Maddox wing test and digit symbol substitution test
Analgesia | 1, 2, 3, 4, 5, 6, 8, 10, 12 hours after the administration of tramadol
  The analgesic effect of tramadol will be evaluated using the cold pressor test. Briefly, the subject's hand is immersed into ice-cold water of + 4° C up to the wrist. The subject is told to keep his or her hand in the water and to report when the cold sensation becomes painful. Cold pain threshold is defined as the latency from the immersion of the hand to the subject's first report of pain. Cold pain intensity is assessed at 30 s intervals following immersion of the hand in cold water for up to 60s . A verbal numerical rating scale of 0-100 will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Intensive Care, Emergency Care and Pain Medicine, Turku University and Turku University Hospital, Turku, Finland